CLINICAL TRIAL: NCT00307879
Title: Phase 2 MAGIC Cell (Myocardial Regeneration and Angiogenesis in Myocardial Infarction With G-CSF and Intra-Coronary Stem Cell Infusion) Trial
Brief Title: Myocardial Regeneration and Angiogenesis in Myocardial Infarction With G-CSF and Intra-Coronary Stem Cell Infusion
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUH-MAGIC1
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2006-03-28 (Estimated); Status verified 2004-03

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; revascularization; granulocyte colony stimulating factor (G-CSF)
MeSH Terms: conditions — Myocardial Infarction

INTERVENTIONS:
Drug: Drug: G-CSF (Dong-A pharmaceutical, Seoul, Korea)
Procedure: collection of mobilized peripheral blood stem cells
Procedure: Intracoronary infusion of mobilized cells

SUMMARY:
This trial was performed to evaluate the safety and the efficacy of G-CSF based stem cell therapy in patients with AMI. MAGIC Cell-1 trial enrolled patients with acute and old myocardial infarction, and had two groups of cell infusion, and G-CSF alone. MAGIC Cell-2 trial enrolled patients with acute myocardial infarction presented within 12 hours after onset of chest pain who underwent successful primary PCI. We randomized patients into the G-CSF group and the control group.

DETAILED DESCRIPTION:
We compared intra-coronary infusion of the mobilized PBSCs with G-CSF (n=10) and mobilization alone with G-CSF (n=10) in patients with myocardial infarction in MAGIC Cell -1 trial and G-CSF alone (n=6) and control (n=6) in MAGIC Cell-2 trial.

This study was a randomized, controlled phase II clinical trial. The Institutional Review Board of Seoul National University Hospital approved the study protocol. The informed written consents were obtained from patients after explaining the procedure and risk.

This study consisted of 2 sub-studies; MAGIC Cell (Myocardial Regeneration and Angiogenesis in Myocardial Infarction with G-CSF and Intra-Coronary Stem Cell Infusion)-1 and 2 trial.

In brief, MAGIC Cell-1 trial enrolled patients with acute and old myocardial infarction, and had two groups of cell infusion, and G-CSF alone. PBSCs were mobilized by daily subcutaneous injections of G-CSF (Dong-A pharmaceutical, Seoul, Korea) with 10 g/kg body weight for four days before percutaneous coronary intervention (PCI). After completion of G-CSF injection, all patients underwent PCI and implantation of stents for the culprit lesion of infarct related artery. Immediately after PCI, patients in the cell infusion group received intra-coronary infusion of the collected PBSC, which were mobilized and collected before PCI. The enrollment of patients to MAGIC Cell-1 trial was terminated prematurely due to potential adverse reaction of increased restenosis. However, follow up of the enrolled patients were completed until 1 year as scheduled. MAGIC Cell-2 trial enrolled patients with acute myocardial infarction presented within 12 hours after onset of chest pain who underwent successful primary PCI. We randomized patients into the G-CSF group and the control group. The patients in the G-CSF group received G-CSF of 10 g/kg body weight for four days at least 24hours after primary PCI. The enrollment of patients to MAGIC Cell-2 trial was also terminated prematurely due to potential adverse reaction of increased restenosis reported in MAGIC Cell-1 trial. However, follow up of the enrolled patients were also completed until 1 year as scheduled

ELIGIBILITY:
Inclusion Criteria:

* MAGIC Cell-1 trial enrolled patients with acute and old myocardial infarction
* MAGIC Cell-2 trial enrolled patients with acute myocardial infarction presented within 12 hours after onset of chest pain who underwent successful primary PCI.

Exclusion Criteria:

* Persistent severe heart failure (above Killip class II or LVEF < 25 %)
* Uncontrolled myocardial ischemia or ventricular tachycardia
* Culprit lesion of infarct related artery not feasible for PCI or unsuccessful PCI
* Age > 75 years
* Malignancy
* Serious current infection or hematologic disease
* Life expectancy under one year.

Ages: 0 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2004-03; Study Completion 2005-02

PRIMARY OUTCOMES:
the change in left ventricular ejection fraction, measured by SPECT, echocardiography

SECONDARY OUTCOMES:
changes in left ventricular volume by SPECT, echocardiography
the development of major adverse cardiac events

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, MD, Principal Investigator — Associated Professor of Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Yon-Gon Dong, Chongno-Gu, Seoul, Seoul, South Korea

REFERENCES:
- [Result] Kang HJ, Kim HS, Zhang SY, Park KW, Cho HJ, Koo BK, Kim YJ, Soo Lee D, Sohn DW, Han KS, Oh BH, Lee MM, Park YB. Effects of intracoronary infusion of peripheral blood stem-cells mobilised with granulocyte-colony stimulating factor on left ventricular systolic function and restenosis after coronary stenting in myocardial infarction: the MAGIC cell randomised clinical trial. Lancet. 2004 Mar 6;363(9411):751-6. doi: 10.1016/S0140-6736(04)15689-4. PMID 15016484